CLINICAL TRIAL: NCT01672827
Title: A Study to Evaluate the Effectiveness of an Electronic Training Program for Orienting and Interpreting [18F]Flutemetamol Positron Emission Tomography (PET) Images.
Brief Title: Effectiveness of an Electronic Training Program for Orienting and Interpreting [18F]Flutemetamol Positron Emission Tomography (PET) Images
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: GE-067-021
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Positron Emission Tomography (PET); PET Images
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — flutemetamol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]Flutemetamol (Experimental)
  Interventions: Drug: [18F]Flutemetamol

INTERVENTIONS:
Drug: [18F]Flutemetamol — No drug is administered in this intervention. These are scanned images being reviewed, previously acquired in various GE-067 studies.
  Other Names: Flutemetamol

SUMMARY:
To Evaluate the Effectiveness of an Electronic Training Program for Orienting and Interpreting [18F]flutemetamol Positron Emission Tomography (PET) Images.

ELIGIBILITY:
Inclusion Criteria:

* Subject received a dose of Flutemetamol F 18 Injection ranging from approximately 185 MBq to approximately 370 MBq.
* The subject was classified as one of the following:

  1. End-of-life subject who expired and underwent brain autopsy, with histochemical (HC) confirmation of brain amyloid status.
  2. Subject with known/suspected normal pressure hydrocephalus (NPH) who underwent brain biopsy, with HC confirmation of brain amyloid status.
  3. Elderly healthy volunteer (age ≥55).
  4. Young healthy volunteer (age ≤40).
  5. Subject with probable Alzheimer Disease (pAD).
  6. Subject with amnestic Mild Cognitive Impairment (aMCI).

Exclusion Criteria:

* Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, MD, Study Chair — GE Healthcare

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study examined brain PET scans from 276 subjects previously acquired form various GE Healthcare studies (GE-067. The study did not enroll the blinded image Readers.
Groups:
- [18F]Flutemetamol: No subjects were dosed for this study. Product was used in scans previously acquired in various GE-067 studies. This study was designed to show the PET Image Interpretations among investigators. The study did not enroll the blinded image Readers.
Period: Overall Study
Arm/Group | [18F]Flutemetamol
Started | 276
Completed | 276
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- [18F]Flutemetamol: No subjects were dosed for this study. Product was used in scans previously acquired in various GE-067 studies. This study was designed to evaluate the effectiveness of an electronic training program for orienting and interpreting Flutemetamol Positive Emission Tomography (PET) Images.
Arm/Group | [18F]Flutemetamol
Number analyzed (Participants) | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 81
  >=65 years | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 140
Region of Enrollment [Number; unit: participants]
  United States | 118
  Belgium | 66
  Denmark | 12
  Finland | 37
  Japan | 16
  Sweden | 3
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Summary of Sensitivity of the Blinded Visual PET Image Interpretations Without Anatomic Images.
Description: Statistical analysis of summary of the blinded visual PET Image Interpretations without Anatomic Images. This data consists of image interpretations by 5 Readers and No subjects were dosed in this study. These Readers examined the PET images for evidence of amyloid plaque.
Time Frame: Post flutemetamol administration
Population: Number of Blinded visual PET Image Interpretations from Readers 1-5. These Readers provided their interpretations without Anatomic Images who had abnormal Standard of Truth (SoT).
Measure: Number (95% Confidence Interval); unit: Percentage (True Positive)
Groups:
- Sensitivity %: Sensitivity of the blinded visual PET Image Interpretations without Anatomic Images.
Arm/Group | Sensitivity %
Number analyzed (Participants) | 51
Percentage (True Positive)
  Reader 1 | 94 [84 to 99]
  Reader 2 | 92 [81 to 98]
  Reader 3 | 90 [79 to 97]
  Reader 4 | 94 [84 to 99]
  Reader 5 | 84 [71 to 93]
  Majority Read | 94 [84 to 99]

2. Secondary Outcome: Inter-Reader Agreement of PET Images Without Anatomic Images
Description: Statistical analysis of Inter-Reader Agreement of PET Images without anatomic Images. This data consists of image interpretations by investigators and No subjects were dosed in this study.
Time Frame: Post Flutemetamol Injection
Measure: Number; unit: Number of inter-reader agreements
Groups:
- Inter-Reader Agreement: Statistical analysis of Inter-Reader Agreement of PET Images without anatomic Images.
Arm/Group | Inter-Reader Agreement
Number analyzed (Participants) | 276
Number of inter-reader agreements
  Reader 1 vs Reader 2 | 248 [73 to 87]
  Reader 1 vs Reader 3 | 257 [.80 to .92]
  Reader 1 vs Reader 4 | 242 [.68 to .83]
  Reader 1 vs Reader 5 | 251 [.75 to .89]
  Reader 2 vs Reader 3 | 255 [.79 to .91]
  Reader 2 vs Reader 4 | 250 [.74 to .88]
  Reader 2 vs Reader 5 | 251 [.75 to .89]
  Reader 3 vs Reader 4 | 253 [.77 to .90]
  Reader 3 vs Reader 5 | 268 [.90 to .98]
  Reader 4 vs Reader 5 | 245 [.71 to .85]
  Readers 1,2,3,4,5 | 223 [.79 to .86]

3. Primary Outcome: Summary of Specificity of Blinded Visual PET Image Interpretations Without Anatomic Images.
Description: Statistical analysis of summary of sensitivity of blinded visual PET image interpretations without anatomic images. This data consists of image interpretations by 5 Readers and No subjects were dosed in this study.These Readers examined the PET images for evidence of amyloid plaque.
Time Frame: Post flutemetamol administration
Population: Number of Blinded visual PET Image Interpretations from Readers 1-5. These Readers provided their interpretations without Anatomic Images who had normal Standard of Truth (SoT).
Measure: Number (95% Confidence Interval); unit: Percentage (True Negative)
Groups:
- Specificity %: Specificity of the blinded visual PET Image Interpretations without Anatomic Images.
Arm/Group | Specificity %
Number analyzed (Participants) | 84
Percentage (True Negative)
  Reader 1 | 79 [68 to 87]
  Reader 2 | 81 [71 to 89]
  Reader 3 | 93 [85 to 97]
  Reader 4 | 77 [67 to 86]
  Reader 5 | 96 [90 to 99]
  Majority Read | 92 [84 to 97]

ADVERSE EVENTS:
Description: No adverse event data collected because no subjects were dosed in this study.
Groups:
- [18F]Flutemetamol: No adverse event data collected because no subjects were dosed in this study , therefore no subjects were at risk.
Arm/Group | [18F]Flutemetamol
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No